CLINICAL TRIAL: NCT01043549
Title: Repetitive Transcranial Magnetic Stimulation of the Posterior Parietal Cortex in Patients Suffering From Gilles de la Tourette Syndrome
Acronym: rTMSPPCGT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lake of efficacy
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C08-46; 2009-A00759-48 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Gilles de la Tourette Syndrome; Tics
Keywords: Gilles de la Tourette syndrome; Tics; Transcranial magnetic stimulation
MeSH Terms: conditions — Tourette Syndrome; Tics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation (Active Comparator): Repetitive transcranial stimulation of the posterior parietal cortex
  Interventions: Device: rTMS
- Sham stimulation (Sham Comparator)
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — Repetitive transcranial stimulation of the posterior parietal cortex
  Arms: Stimulation
Device: Sham rTMS — Repetitive transcranial stimulation of the posterior parietal cortex
  Arms: Sham stimulation

SUMMARY:
Repetitive transcranial stimulation (rTMS) of the posterior parietal cortex will be applied daily over five days in adult Gilles de la Tourette patients. This approach aims at reducing premonitory sensations believed to induce tics. Patients will be randomized to an active or placebo (sham) group in a crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Gilles de la Tourette syndrome as defined by DSM IV-R
* Yale Global Tics Severity Scale (YGTSS) score between 30 et 60
* Premonitory sensations (" urge to move ")
* Affiliated to the French social security regime
* Ability to give informed consent

Exclusion Criteria:

* rTMS : epilepsy, craniotomy scar, pacemaker or neural stimulator, metal implants or foreign bodies, claustrophobia, pregnancy
* Cognitive impairment (MMS ≤ 24/30)
* Axis I disorders according to DSM IV-R : psychosis or history of psychosis, bipolar illness, major depressive disorder, addictions (except to nicotine)
* Impulse control disorders
* Other chronic debilitating illnesses
* Unability to give informed consent
* Participation in another clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Yale global tic severity scale (YTGSS) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hartmann, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Inserm U975, Paris, France